CLINICAL TRIAL: NCT00632034
Title: A Phase I Safety Study Following the Infusion of Expanded Autologous Progeny of an Adult CD34+ Stem Cell Subset to Patients With Recent Tibial Fractures
Brief Title: Stem Cells and Tibial Fractures
Acronym: STIF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HHSC/010; 2006-004521-28 (EudraCT Number)
Record Dates: First submitted 2008-02-29; First posted 2008-03-10 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Tibial Fractures
Keywords: fracture; tibia; stem cell
MeSH Terms: conditions — Tibial Fractures; Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Other: CD34+ haemopoietic stem cells

INTERVENTIONS:
Other: CD34+ haemopoietic stem cells — Expanded subset of CD34+ haemopoietic stem cell. Harvested from pelvic marrow aspiration at Day 0 of study. Undergoes refinement and minimum of 1000 fold expansion over 7 days in a dose escalation regime of a maximum dose of 1,000,000,000 cells in 5 millilitres. Injected at Day 7 via contralateral femoral artery under angiographic guidance. First regime up to 10,000,000 cells, second 100,000,000 cells, final regime maximum of 1,000,000,000 cells.
  Other Names: Omnicyte

SUMMARY:
The aim of this trial is to determine the safety and tolerability of expanded autologous progeny of an adult CD34+ (haemopoietic) stem cell subset when infused directly into the tibial artery of patients with recent tibial fracture. The trial will also seek to determine clinical improvement or deterioration by measurement of clinical parameters such as, length of time to union of the fracture, changes in bone mineral density, improvements in pain scores (VAS), functional ability (TUGT) and IPAQ scores.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed closed tibial fracture on one limb only
* Normal blood count
* Normal coagulation screen
* Life expectancy of at least 12 months
* Ability to give written informed consent

Exclusion Criteria:

* Patients with additional lower limb injuries
* Patients with abnormal lower limb vasculature
* Pregnant or lactating women
* Unexplained abnormal baseline laboratory results
* Males and females who are capable of reproduction and will not take acceptable measures to prevent reproduction during the study
* Subjects who test positive for HTLV, HIV, hepatitis B or hepatitis C, have a chronic inflammatory disease, autoimmune disease or are on chronic immunosuppressive medications
* History of alcohol or drug abuse within 3 months of screening
* Subjects with evidence (clinical, laboratory, or imaging) of cancer or cancer recurrence within the past 5 years (other than non-melanoma skin cancer or in situ cervical carcinoma)
* Currently enrolled in another investigational device or drug trial that has not completed the required follow-up period
* Patients unable to give written informed consent

Ages: 17 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-05 (Estimated); Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
To assess the safety of expanded autologous progeny of an adult CD34+ stem cell subset when introduced into the tibial artery and to determine absence of adverse events at the maximum dose of cells of 1,000,000,000 cells in a dose escalation regime. | 1 year

SECONDARY OUTCOMES:
To assess improvement in bony union as measured by imaging modalities and determine whether there are any significant improvements in early restoration of function as reported by the patients. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sean P.F. Hughes, MS, Principal Investigator — Imperial College London
Locations (1):
- Charing Cross Hospital, London, United Kingdom

REFERENCES:
- [Background] Bianco P, Gehron Robey P. Marrow stromal stem cells. J Clin Invest. 2000 Jun;105(12):1663-8. doi: 10.1172/JCI10413. No abstract available. PMID 10862779
- [Background] Bruder SP, Kraus KH, Goldberg VM, Kadiyala S. The effect of implants loaded with autologous mesenchymal stem cells on the healing of canine segmental bone defects. J Bone Joint Surg Am. 1998 Jul;80(7):985-96. doi: 10.2106/00004623-199807000-00007. PMID 9698003
- [Background] Dickson K, Katzman S, Delgado E, Contreras D. Delayed unions and nonunions of open tibial fractures. Correlation with arteriography results. Clin Orthop Relat Res. 1994 May;(302):189-93. PMID 8168299
- [Background] Dunlop DD, Hughes SL, Edelman P, Singer RM, Chang RW. Impact of joint impairment on disability-specific domains at four years. J Clin Epidemiol. 1998 Dec;51(12):1253-61. doi: 10.1016/s0895-4356(98)00128-0. PMID 10086817
- [Background] Friedlaender GE, Perry CR, Cole JD, Cook SD, Cierny G, Muschler GF, Zych GA, Calhoun JH, LaForte AJ, Yin S. Osteogenic protein-1 (bone morphogenetic protein-7) in the treatment of tibial nonunions. J Bone Joint Surg Am. 2001;83-A Suppl 1(Pt 2):S151-8. PMID 11314793
- [Background] Grazier KL, Holbrook TL, Kelsey JL, Stauffer RN. The frequency of occurrence, impact, and cost of musculoskeletal conditions in the United States. American Academy of orthopaedic Surgeons Chicago IL, USA. 1984
- [Background] Heppenstall RB, Brighton CT, Esterhai JL Jr, Muller G. Prognostic factors in nonunion of the tibia: an evaluation of 185 cases treated with constant direct current. J Trauma. 1984 Sep;24(9):790-5. PMID 6332920
- [Background] NICOLL EA. FRACTURES OF THE TIBIAL SHAFT. A SURVEY OF 705 CASES. J Bone Joint Surg Br. 1964 Aug;46:373-87. No abstract available. PMID 14216447
- [Background] Kadiyala S, Young RG, Thiede MA, Bruder SP. Culture expanded canine mesenchymal stem cells possess osteochondrogenic potential in vivo and in vitro. Cell Transplant. 1997 Mar-Apr;6(2):125-34. doi: 10.1177/096368979700600206. PMID 9142444
- [Background] KUNTSCHER G. [Medullary nailing of fractures of tibial shaft]. Langenbecks Arch Klin Chir Ver Dtsch Z Chir. 1953;276:217-27. No abstract available. Undetermined Language. PMID 13143788
- [Background] Lee EH, Hui JH. The potential of stem cells in orthopaedic surgery. J Bone Joint Surg Br. 2006 Jul;88(7):841-51. doi: 10.1302/0301-620X.88B7.17305. No abstract available. PMID 16798982
- [Background] Lieberman JR, Daluiski A, Einhorn TA. The role of growth factors in the repair of bone. Biology and clinical applications. J Bone Joint Surg Am. 2002 Jun;84(6):1032-44. doi: 10.2106/00004623-200206000-00022. No abstract available. PMID 12063342
- [Background] Singer BR, McLauchlan GJ, Robinson CM, Christie J. Epidemiology of fractures in 15,000 adults: the influence of age and gender. J Bone Joint Surg Br. 1998 Mar;80(2):243-8. doi: 10.1302/0301-620x.80b2.7762. PMID 9546453
- [Background] Vats A, Tolley NS, Buttery LD, Polak JM. The stem cell in orthopaedic surgery. J Bone Joint Surg Br. 2004 Mar;86(2):159-64. doi: 10.1302/0301-620x.86b2.14756. No abstract available. PMID 15046426